CLINICAL TRIAL: NCT00223249
Title: A Randomized, Double-Blind, Placebo-Controlled Add-On Trial of Quetiapine in Patients With Bipolar Disorder and Alcohol Abuse/ Dependence.
Brief Title: Quetiapine in Patients With Bipolar and Alcohol Abuse/Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRUSQUET0233
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Bipolar Disorder; Alcohol Abuse/Dependence
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine (Active Comparator): Quetiapine
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator): Inactive ingredient matching the active medication in appearance
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
The abuse of alcohol is especially common in people with bipolar disorder. However, very little is known about the pharmacotherapy of people with both bipolar disorder and alcohol abuse/dependence. The purpose of this study is to determine if alcohol use and cravings are decreased with quetiapine add-on therapy compared to placebo and to determine if quetiapine add-on therapy is associated with greater improvement in mood, impulsivity, functioning and decreased alcohol use than placebo.

DETAILED DESCRIPTION:
Experimental: After obtaining informed consent, 100 patients with bipolar I, or II disorders and alcohol abuse/dependence confirmed by a structured clinical interview (SCID) will be enrolled. from referral sources in the community we have developed over the past 3 years. A medical history and physical examination, including an eye exam with an ophthalmoscope, will also be performed at baseline to rule out serious medical illnesses and cataracts. Baseline labs including a liver panel and CBC will be obtained. Women of child-bearing potential will be given a urine pregnancy test. Baseline measures of psychiatric symptoms will be assessed with the HRSD, YMRS, and Barratt Impulsiveness Scale. Alcohol cravings will be assessed with the Obsessive Compulsive Drinking Scale (OCDS). Alcohol use including number of drinks/2 weeks, days used in the past two weeks, and days of heavy use will be obtained as will a urine drug/alcohol screen. Alcohol use and cravings will also be recorded throughout the study. Side-effects will be assessed with a general side effects scale, the Abnormal Involuntary Movement Scale (AIMS), Simpson-Angus Scale (SAS), and Barnes Akathesia Rating Scale (BARS). GGT levels will also be repeated at weeks 6 and 12. The subjects will be randomized and receive quetiapine or identical appearing placebo add-on therapy in a double-blind fashion for 12 weeks. Subjects will return every two weeks for reevaluation with the above outcome measures and for upward titration of study drug. All subjects will be given the option of receiving open-label quetiapine for an additional 4 weeks (with continuing assessment of mood and alcohol use/cravings every 2 weeks) at the end of the study or discontinuing medication.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I or II
* Ages 18-70

Exclusion Criteria:

* Life threatening medical condition causing participation in the study hazardous
* Alcohol abuse within the past 2 weeks
* History of cataracts or likely cataracts on baseline eye exam
* History of hepatic cirrhosis or AST or ALT more than three times normal limit
* Current active suicidal or homicidal ideation
* History of allergic reaction, poor response or intolerable side effects to quetiapine
* Antipsychotic use within 7 days of beginning quetiapine therapy
* Mental retardation, dementia or other severe cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2002-11; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Number of Standard Drinks | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, Ph.D., M.D., Principal Investigator — The UT Southwestern Medical Center at Dallas
Locations (1):
- The UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Brown ES, Garza M, Carmody TJ. A randomized, double-blind, placebo-controlled add-on trial of quetiapine in outpatients with bipolar disorder and alcohol use disorders. J Clin Psychiatry. 2008 May;69(5):701-5. doi: 10.4088/jcp.v69n0502. PMID 18312058